CLINICAL TRIAL: NCT01155024
Title: Clinical Evaluation of Direct Manufactured Prosthetic Sockets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio Willow Wood (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-08-10700-V1
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-12

CONDITIONS: Amputation
Keywords: Lower extremity amputation; Prosthetic Sockets; Direct Manufactured (DM)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Socket First, then DM Socket (Other): Initial fitting of a traditional diagnostic prosthetic socket in first intervention period and initial fitting of a direct manufactured prosthetic socket in the second intervention period
  Interventions: Device: Traditional fabricated prosthetic socket; Device: Direct manufactured (DM) prosthetic socket
- DM Socket First, then Traditional Socket (Other): Initial fitting of a direct manufactured prosthetic socket in first intervention period and initial fitting of a traditional diagnostic prosthetic socket in the second intervention period
  Interventions: Device: Traditional fabricated prosthetic socket; Device: Direct manufactured (DM) prosthetic socket

INTERVENTIONS:
Device: Traditional fabricated prosthetic socket — A prosthetic socket constructed utilizing traditional techniques. This intervention is a control and the basis for comparison.
  Other Names: Rectified prosthetic socket
Device: Direct manufactured (DM) prosthetic socket — A prosthetic socket constructed from direct manufacturing technique. The socket will be tested under both diagnostic and definitive environments. Diagnostic testing will span several hours (4-6 hours) and definitive testing will span several months (3-6 months)

SUMMARY:
The purpose of this study is to evaluate a new prosthetic socket construction technique in order to improve the quality of care to lower extremity amputees.

DETAILED DESCRIPTION:
Many members of the Armed Forces and civilians are in need of prosthetic devices due to amputations resulting from gunshots, bombings, vehicular accidents, and other traumas. As the number of amputees increase at a high rate, the limited number of certified prosthetists is finding it harder to satisfy the patient demand. Therefore, the overall goal is to provide the Orthopedic & Prosthetic (O&P) industry with a tool that accommodates the increasing prosthetist to patient ratio and still provide acceptable product quality.

The practice of creating prosthetic sockets by the plaster-casting of amputees' residual limbs has been around for decades but continues to be the most commonly used method for the shape capture, modification and fabrication of prosthetic sockets. Using this traditional plaster-casting approach has many limitations that can now be overcome through the use of technology.

With the advancing developments in Computer Aided Design (CAD) and Computer Aided Manufacturing (CAM) technologies over the past ten years, it is now possible to completely replace the plaster-casting approach with handheld, portable scanners.

While this current CAD/CAM approach certainly creates substantial efficiencies in the clinical aspects of creating the prosthetic socket, the actual manufacturing of the prosthetic device continues to rely on the use of a positive model and a lengthy manual fabrication process.

The continuing development of direct manufacturing technologies may serve as the final piece in the effective utilization of CAD/CAM in the care of prosthetic and orthotic patients. Direct manufacturing provides a means to quantify alterations and accurately reproduce prosthetic sockets. Additionally, direct manufacturing has the potential to reduce time, cost, and waste, as a result improve the quality and care ability to patients.

This study will compare two fabrication techniques for diagnostic and definitive sockets: manually fabricated (positive model technique) and direct manufactured (experimental).

ELIGIBILITY:
Inclusion Criteria:

* Be a lower extremity amputee longer than one year
* Be a consenting adult (at least 18 years or age or older)
* Albe to ambulate in current prosthesis without an aid (can, crutches or walker) for 30 minutes without rest
* Currently using a liner with prosthesis
* Be available during regular business hours for appointments

Exclusion Criteria:

* An inability to give informed consent
* Presence of any sores, lacerations or rashes on the residual limb
* Impaired contra lateral foot
* Poor distal sensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Colvin, M.S., Principal Investigator — Ohio Willow Wood
Locations (1):
- Ohio Willow Wood, Mount Sterling, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between March 2011 and June 2011
Pre-assignment Details: 10 participants recruited; 10 screened, 0 excluded
Groups:
- Traditional Socket: Initial fitting of a traditional diagnostic prosthetic socket
- Direct Manufactured Socket: Initial fitting of a direct manufactured prosthetic socket
Period: First Socket Intervention Fitting
Arm/Group | Traditional Socket | Direct Manufactured Socket
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Socket Intervention Fitting
Arm/Group | Traditional Socket | Direct Manufactured Socket
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Direct Manufactured Socket 3 Month Trial
Arm/Group | Traditional Socket | Direct Manufactured Socket
Started | 0 | 10
Completed | 0 | 4
Not Completed | 0 | 6
Not completed — Experienced inferior suspension system | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive the traditional diagnostic prosthetic socket first and the direct manufactured prosthetic socket first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Weight [Mean (Standard Deviation); unit: kg] | 106 (24.7)
Number of years participant has worn a Prosthesis [Mean (Standard Deviation); unit: years] — Total number of years the participant has worn a lower limb prosthesis
  years | 13.4 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Hanspal Socket Comfort Score (SCS) After Initial Socket Fitting
Description: The Hanspal SCS assesses participant socket comfort on a continuous scale from 0 (most uncomfortable) to 10 (most comfortable)
Time Frame: Within the first 4-6 hrs
Population: Per protocol analysis including all consented participants
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Traditional Socket: Traditional diagnostic prosthetic socket fitted using typical fitting techniques in either the first intervention period or second intervention period.
- Direct Manufactured Socket: Direct manufactured prosthetic socket fitted using typical fitting techniques in either the first intervention period or second intervention period.
Arm/Group | Traditional Socket | Direct Manufactured Socket
Number analyzed (Participants) | 10 | 10
score on scale | 9 (0.82) | 8.7 (0.82)
Statistical Analysis 1: Comparison: Traditional Socket vs Direct Manufactured Socket; Alpha level of 0.05; Test type: Non-Inferiority or Equivalence — 10 participants required to detect one value change in rating for the SCS scale, with 80% power; p > 0.4, t-test, 2 sided — Two-Sided

2. Secondary Outcome: Participant Socket Preference After Initial Fitting
Description: Number of participants indicating socket preference after initial fitting of both socket interventions
Time Frame: Within the first 4-6 hours
Population: Total number of participants completing period for both study interventions.
Measure: Number; unit: participants
Groups:
- Socket Preference: Participant's indicated preference of socket type (preferred traditional socket, preferred direct manufactured socket, or no preference/difference)
Arm/Group | Socket Preference
Number analyzed (Participants) | 10
participants
  Preferred Traditional Socket | 2
  Preferred Direct Manufactured Socket | 0
  No Preference/Difference | 8

3. Secondary Outcome: Participant Socket Preference After 3 Months Usage of the Direct Manufactured Socket
Description: Number of participants indicating socket preference after 3 months usage of the direct manufactured prosthetic socket. Comparisons made to their previous traditional definitive prosthetic socket
Time Frame: 3 months
Population: Total number of participants completing the period (3 months usage of direct manufactured socket) and participants classified as 'Withdrawal by participant'. Analysis does not include participants who prematurely withdrew for reasons unrelated to the direct manufactured socket intervention.
Measure: Number; unit: participants
Arm/Group | Socket Preference
Number analyzed (Participants) | 6
participants
  Preferred Traditional Socket | 2
  Preferred Direct Manufactured Socket | 4
  No Preference/Difference | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Traditional Socket | Direct Manufactured Socket
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Early termination by four participants for reasons unrelated to the interventions lead to smaller numbers completing the 3 month trial period for the direct manufactured socket.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No